CLINICAL TRIAL: NCT00471926
Title: Diabetes Quality Improvement Program on Diabetes Case Management Program 2001
Acronym: DQIP-DCMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Other Study IDs: DMR96-IRB-41
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In order to assess more completely the levels of diabetes care delivered in Taiwan, we now have nationally standardized performance measures that can evaluate quality of diabetes care accurately and reliably. These performance measures were seriously reviewed and discussed in the aspects of their practicability, feasibility and compliancy, through a series of nation-wide consensus meetings by a number of multidisciplinary professionals of Taiwan Diabetes Care Teams ( TDCTs ), before delivering into the clinical settings ( 10 ).

Conceptually, these measures will enhance uptake of research into practice and may ultimately improve diabetes care and clinical outcomes. Along with the serial developments mentioned above, the BNHI ( the sole healthcare insurance organization in Taiwan ) has been fully involved, from the very beginning, in the formation and development of these performance measures which have totally been included in the development of the Diabetes Case Management Program ( DCMP ) 2001 later on. The DCMP 2001 is a unique program that has been delivered into the nation-wide clinical practices since Dec. 2001 in Taiwan. It has linked the quality of diabetes care to the monthly income ( reimbursed from BNHI ) of the registered clinical diabetes educators ( i.e., physicians, nurses and dietitians ) for enhancing and assuring the complete implementation of these performance measures in diabetes care. It has been recognized that a consensus on measures at national level could provide a method for assessing care within and across healthcare settings while providing a meaningful mechanism for quality improvement. In this proposal, we are going to develop the Diabetes Quality Improvement Program ( DQIP ) based on the DCMP 2001 in Taiwan.

Initially, we are going to establish the continuous diabetes quality monitoring system and then to evaluate the (1) the lifestyles and eating habits and dietary compositions in type 2 diabetes mellitus (2)The relationships between lifestyles and eating habits and dietary compositions in diabesity.

DETAILED DESCRIPTION:
Diabetes is now a global epidemic; it is the fourth or fifth leading cause of death in most developed and newly industrialized countries. People with diabetes mean a long-term condition that deserves effective and efficient care throughout their lives. Complications caused by diabetes, such as coronary artery and peripheral vascular diseases, stroke, diabetic neuropathy, amputations, renal failure and blindness are resulting in increasing disability, reduced life expectancy and, even more apprehensive, enormous healthcare related expense for virtually every society ( 1, 2 ). Diabetes is certainly one of the most challenging health issues in the 21st century.

The most recent epidemiological data suggested that the diabetes population in Taiwan has reached one million ( 3 ). People with diabetes using the healthcare insurance regularly for their diabetes care, however, were only 60 % of total diabetes population. Nevertheless, this 60 % of Taiwan diabetes population had already consumed more than 12 % of total national annual healthcare expenditure in taking care of them. In fact, this diabetes population was merely one- forties of Taiwan population as a whole. Even the worst thing was that more than 60 % of the whole yearly healthcare budget for taking care of diabetes had gone into the treatment of diabetes-related complications ( 4,5 ). We have recently learned from some of the prevention trials, such as the Diabetes Control and Complications Trial ( DCCT ) in type 1 diabetes and the United Kingdom Prospective Diabetes Study ( UKPDS ) in type 2 diabetes, that effective and adequate performance of metabolic and blood pressure control in patients with diabetes would be able to delay or even prevent the diabetes-related complications ( 6-8 ). These interventions, if broadly implemented, would help to improve the living quality of diabetes patients, and as well as to consequently make the biggest gain out of healthcare expenditure ( 9 ). In order to assess more completely the levels of diabetes care delivered in Taiwan, we now have nationally standardized performance measures that can evaluate quality of diabetes care accurately and reliably. These performance measures were seriously reviewed and discussed in the aspects of their practicability, feasibility and compliancy, through a series of nation-wide consensus meetings by a number of multidisciplinary professionals of Taiwan Diabetes Care Teams ( TDCTs ), before delivering into the clinical settings ( 10 ).

Conceptually, these measures will enhance uptake of research into practice and may ultimately improve diabetes care and clinical outcomes. Along with the serial developments mentioned above, the BNHI ( the sole healthcare insurance organization in Taiwan ) has been fully involved, from the very beginning, in the formation and development of these performance measures which have totally been included in the development of the Diabetes Case Management Program ( DCMP ) 2001 later on. The DCMP 2001 is a unique program that has been delivered into the nation-wide clinical practices since Dec. 2001 in Taiwan. It has linked the quality of diabetes care to the monthly income ( reimbursed from BNHI ) of the registered clinical diabetes educators ( i.e., physicians, nurses and dietitians ) for enhancing and assuring the complete implementation of these performance measures in diabetes care. It has been recognized that a consensus on measures at national level could provide a method for assessing care within and across healthcare settings while providing a meaningful mechanism for quality improvement. In this proposal, we are going to develop the Diabetes Quality Improvement Program ( DQIP ) based on the DCMP 2001 in Taiwan.

Initially, we are going to establish the continuous diabetes quality monitoring system and then to evaluate the (1) the lifestyles and eating habits and dietary compositions in type 2 diabetes mellitus (2)The relationships between lifestyles and eating habits and dietary compositions in diabesity.

ELIGIBILITY:
Inclusion Criteria:

* All of Diabetes Cases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2007-04; Study Completion 2008-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fuh, MD,DMSci, Principal Investigator — mmtfuh@www.cmuh.org.tw
Locations (1):
- Martin M-T Fuh, Taichung, Taiwan